CLINICAL TRIAL: NCT04994912
Title: Title of Study: A First-in-Human, Phase 1, Randomized, Double-Blind, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of EI-001 in Healthy Volunteers
Brief Title: First in Human Study of EI-001 Monoclonal Antibody in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elixiron Immunotherapeutics (Hong Kong) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EI-001-101
Record Dates: First submitted 2021-07-19; First posted 2021-08-06 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy
MeSH Terms: interventions — BL-EI001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EI-001 (Experimental): IV infusion
  Interventions: Drug: EI-001
- Placebo (Placebo Comparator): IV infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: EI-001 — EI-001 IV infusion
  Arms: EI-001
Other: Placebo — Placebo IV infusion
  Arms: Placebo

SUMMARY:
A First-in-Human, Phase 1, Randomized, Double-Blind, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of EI-001 in Healthy Volunteers.

DETAILED DESCRIPTION:
To assess the safety and tolerability of single ascending intravenous (IV) doses of EI-001 in healthy volunteers

To assess the pharmacokinetics (PK) of single ascending IV doses of EI-001 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female 18 to ≤ 55 years old at the time of consent.
2. Healthy on the basis of physical examination, medical history, vital signs, laboratory values and 12-lead ECG performed at Screening. The participant may be included only if the investigator judges any abnormalities or deviations from normal to be not clinically significant.

Exclusion Criteria:

1. Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the Investigator's (or delegate's) opinion, may require treatment or render the participant unlikely to fully complete the study, or any condition that presents undue risk from the IP or procedures or interfere with study assessments.
2. Have received any IP within 30 days or 5 half-lives prior to Screening (4 months if the previous drug was a new chemical entity), whichever is longer.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
safety assessment | Day 1
  to assess blood pressure
safety assessment | Day 1
  to assess heart rate
safety assessment | Day 1
  to assess respiratory rate

SECONDARY OUTCOMES:
PK assessment | Day 1
  To assess Maximum observed concentration (Cmax)
PK assessment | Day 1
  To assess time to maximum observed drug concentration (Tmax)
PK assessment | Day 1
  to assess AUC from time zero to the last measurable concentration (AUC0-t)

CONTACTS AND LOCATIONS:
Locations (2):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia
- Huashan Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No